CLINICAL TRIAL: NCT06010771
Title: The Effect of Listening to Stories and Watching Cartoon Film on Pain in the Aspiration Process in Playing Age Children Receiving Palliative Care: A Randomized Controlled Trial
Brief Title: The Effect of Listening to Stories and Watching Cartoon Film on Pain in the Aspiration Process in Children Receiving Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gamze Akay (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, Gamze Akay, Lecturer, Artvin Coruh University
Organization: Artvin Coruh University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pediatric Nursing
Record Dates: First submitted 2023-06-30; First posted 2023-08-25 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Aspiration; Syndrome
Keywords: Palliative care; Children; Listening to Stories; Watching Cartoon Film; Pain
MeSH Terms: conditions — Syndrome; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine aspiration will be applied to the control group. No action will be taken.
- Experimental Group (Experimental): During the aspiration process, the experimental group will listen to fairy tales and watch cartoons.
  Interventions: Other: Listening to fairy tales; Other: Watching Cartoon Film

INTERVENTIONS:
Other: Listening to fairy tales — Fairy tales by children will be chosen by child psychologists. Tales will be read to the children by the researcher. The researcher has a fairy tale therapy certificate. The tale reading will start 5 minutes before the aspiration process and will continue throughout the aspiration process. Tales will be read to children every other day. This process will continue for 3 weeks.
  Arms: Experimental Group
Other: Watching Cartoon Film — The cartoons that children will watch will be preferred by child psychologists. Children will be watched cartoons with the help of tablets. Watching cartoons will start 5 minutes before the aspiration process and will continue throughout the aspiration process. Children will be shown cartoons every other day. This process will continue for 3 weeks.
  Arms: Experimental Group

SUMMARY:
The aim of this study is to determine the effect of listening to fairy tales and watching cartoons on pain in the aspiration process in play-age children receiving palliative care.

DETAILED DESCRIPTION:
15 voluntary children with receiving palliative care, aged between 1-3 years will be randomly divided into two groups: fairy tale group and cartoon group. Interventions will be applied for 3 weeks, 1 times a day (16 sessions). No intervention will be applied to both groups besides fairy tale or cartoon intervention. The children will be assessed before, during and after. PAIN DUE TO ASPIRATION PROCEDURE will be evaluated using the FLACC Pain Scale. In addition, the heart rate, respiration, blood pressure, tidal volume and fever values of the children will be measured with the help of a bedside monitor.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 1-3 age group
* Being in the palliative care service for at least 3 months
* Receiving inpatient treatment in the pediatric palliative care service
* Absence of visual and hearing anomalies
* No other chronic disease
* Having a tracheostomy

Exclusion Criteria:

* The family's desire to leave research.
* Deterioration of the child's condition
* The child's diagnosis of an additional chronic disease

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
Patient Identification Form | baseline
  In this form, there are questions about the child's age, gender, diagnosis of the disease, length of stay, and how long ago she received the current diagnosis.
Physiological Parameter Record Form | baseline and up to 4 weeks
  In this form, there are records of all physiological parameters including pulse and respiratory rate, body temperature, blood pressure, SpO2, tidal volume, and peak heart rate. If the value of each parameter is higher than the normal values, it indicates the presence of abnormal condition.
  Pulse normal value range: 80-130/ Minute Blood pressure normal value range:92-44 mmHg Respiratory rate normal value range: 16-22/ Minute Body temperature normal value range: 36,4-38 degree SpO2 normal value range: %96-98 Tidal volume normal value range: 6-10 ml/kg
FLACC Pain Scale | baseline and up to 4 weeks
  FLACC has reliability and validity to determine observational pain of children aged between 3 and 18 years during the medical procedures. This scale is preferred due to its implicity of application among children. It has five categories of behavior to rate pain, namely, facial expression, leg movement, activity, cry, and consolability. The scores of each category are between 0 and 2. The total scores can range from 0 to 10, defined as mild (1-3), moderate (4-6), and severe (7-10). The higher the score, the greater the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze AKAY, 1, Principal Investigator — Artvin Coruh University
Locations (1):
- Erzurum City Hospital, Erzurum, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarialioglu A, Kurudirek F, Oluc T. The effect of storybook reading on children's preoperative fear and anxiety levels: A randomized controlled study. Child Care Health Dev. 2023 Sep;49(5):906-913. doi: 10.1111/cch.13100. Epub 2023 Feb 8. PMID 36735635
- See also: A randomized controlled study — http://pubmed.ncbi.nlm.nih.gov/36735635/